CLINICAL TRIAL: NCT07126795
Title: Magnesium Sulfate for Adjuvant Analgesia in Pediatric Burn Dressing Changes: a Pilot Study
Brief Title: Magnesium Sulfate in Pediatric Burn Dressing Changes
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Joseph Resch, PICU Physician, Assistant Professor, Associate Program Director, PCCM Fellowship, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HCMC Pediatric Burn Study
Record Dates: First submitted 2025-08-04; First posted 2025-08-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Burns
Keywords: magnesium sulfate; pediatrics; burn; analgesia; sedation; burn dressing change
MeSH Terms: conditions — Burns; Agnosia | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate Arm (Experimental): Pediatric Burn Patients receiving Ketamine as primary agent for sedated dressing changes, randomized (max 5 randomizations) to either study intervention (Magnesium sulfate) or placebo (Normal saline)
  Interventions: Drug: magnesium sulfate
- Normal Saline Placebo Arm (Placebo Comparator): Placebo
  Interventions: Drug: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: magnesium sulfate — IV Magnesium Sulfate 50 mg/kg (max 2 grams) over 20 minutes given immediately prior to initiation of daily sedated dressing change
  Arms: Magnesium Sulfate Arm
Drug: Normal Saline (0.9% NaCl) — Normal Saline given in equivalent volume as study drug over 20 minutes, immediately prior to initiation of sedated dressing change
  Arms: Normal Saline Placebo Arm

SUMMARY:
Prospective feasibility trial utilizing adjuvant magnesium sulfate for analgesia/sedation during pediatric sedated burn dressing changes, which is ultimately hypothesized to decrease ketamine and/or sedative requirements.

DETAILED DESCRIPTION:
Pediatric patients (n=10) suffering severe burn, admitted to the burn unit at Hennepin County Medical Center (Minneapolis, MN) meeting specific inclusion/exclusion criteria will be randomized daily to either intravenous magnesium sulfate (50 mg/kg, max 2 g) or placebo (normal saline) for up to 5 sedated burn dressing changes. Primary aims will be to evaluate safety/feasibility to guide a future larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* < 18 years old at time of randomization completion
* admission to HCMC Burn Unit
* Projected multi-day sedated dressing change requirement
* Intention for IV Ketamine as primary analgosedative agent

Exclusion Criteria:

* age < 3 years (may lower pending FDA discussions)
* Evidence of hypermagnesemia - pre-study serum Mg2+ level > 2.5 mg/dL
* Evidence of renal dysfunction - serum Cr level > 1.5x hospital upper limit normal for age
* Presence of neuromuscular disease (specifically myasthenia gravis), underlying bradyarrhythmia or heart block
* Bronchospastic disease (asthma, reactive airway disease) which requires continuous magnesium sulfate infusion
* Active prescription of a calcium channel blocker (amlodipine, isradipine, nicardipine, nifedipine, clevidipine, diltiazem, verapamil), cardiac glycoside (digoxin), parenteral nutrition or an infusion for hemodynamic support (epinephrine, norepinephrine, dopamine, dobutamine, milrinone, etc)
* Known allergy or reaction to magnesium sulfate, aluminum, or a component of the formulation
* Presence of invasive mechanical ventilation
* Anticipation of skin grafting within 5 days of study eligibility
* Anyone whom child protective services are consulted
* Any investigational drug use within 30 days prior to enrollment
* Pregnant or lactating females
* Anyone whom in the opinion of the investigator is at higher than anticipated risk of harm or inability to adhere to protocol
* Patients who choose to opt out of research

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Severe Adverse Events | Through Study Completion, Approximately 1 year
  Frequency of severe adverse events
Protocol Deviations | Through Study Completion, Approximately 1 year
  Number of Protocol Deviations
Consent Rate | Through Study Completion, Approximately 1 year
  Consent Rate (%)
Enrollment Effort | Through Study Completion, Approximately 1 year
  Enrollment Effort of Study Personnel (hours)
Study Duration Indicator | Through Study Completion, Approximately 1 year
  Duration to Reach Enrollment Target (months)
Effectiveness of Drug Delivery & Timing | Through Study Completion, Approximately 1 year
  Magnesium Sulfate Completion Timing, Relative to Sedation Start Time (minutes)
Extra Blood Draws | Through Study Completion, Approximately 1 year
  Number of Extra Blood Draws per Patient

SECONDARY OUTCOMES:
Ketamine dosage | Through Study Completion, Approximately 1 year
  Cumulative dose requirement of ketamine during sedated dressing change (mg/kg)
Adverse Events | Through Study Completion, Approximately 1 year
  Specific tracking of adverse events related to Magnesium sulfate and deep sedative agents. General tracking of adverse events. Description of severity and relation to magnesium sulfate.

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No